CLINICAL TRIAL: NCT06842472
Title: A Prospective Phase II Randomized Clinical Trial of PD-L1 Monoclonal Antibody in Combination with Radiation Therapy, with or Without Ursodeoxycholic Acid, in Patients with Recurrent or Metastatic HER2-Negative Breast Cancer
Brief Title: PD-L1 Inhibitor + RT ± Ursodeoxycholic Acid in Recurrent/Metastatic HER2-Neg Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang, Prof, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5137；Approve No.25/004-0004
Record Dates: First submitted 2025-02-12; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ursodeoxycholic Acid; Radiotherapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Adebrelimab (PD-L1 inhibitor) 1200 mg on Day 1, every 3 weeks. Radiotherapy (SBRT) with a dose of 24Gy/3 fractions within 3 weeks after the first immunotherapy dose.
  UDCA 250 mg twice daily, starting 7 days before radiotherapy and continuing for 1 month after radiotherapy completion.
  Interventions: Drug: Ursodeoxycholic Acid (URSO); Radiation: Radiotherapy; Drug: Adebrelimab (PD-L1 inhibitor)
- Control Group (Active Comparator): Adebrelimab 1200 mg on Day 1, every 3 weeks. Radiotherapy (SBRT) with a dose of 24Gy/3 fractions within 3 weeks after the first immunotherapy dose.
  Interventions: Radiation: Radiotherapy; Drug: Adebrelimab (PD-L1 inhibitor)

INTERVENTIONS:
Drug: Ursodeoxycholic Acid (URSO) — UDCA 250 mg twice daily, starting 7 days before radiotherapy and continuing for 1 month after completion.
  Arms: Experimental Group
Radiation: Radiotherapy — Radiotherapy (SBRT) with a dose of 24Gy/3 fractions within 3 weeks after the first immunotherapy dose.
Drug: Adebrelimab (PD-L1 inhibitor) — Adebrelimab (PD-L1 inhibitor) 1200 mg on Day 1, every 3 weeks.

SUMMARY:
Experimental Group Adebrelimab (PD-L1 inhibitor) 1200 mg on Day 1, every 3 weeks. Radiotherapy (Stereotactic Body Radiation Therapy, SBRT) with a dose of 24 Gy/3 fractions within 3 weeks after the first immunotherapy dose.

Ursodeoxycholic Acid (UDCA) 250 mg twice daily, starting 7 days before radiotherapy and continuing for 1 month after radiotherapy completion.

Control Group Adebrelimab 1200 mg on Day 1, every 3 weeks. SBRT with a dose of 24 Gy/3 fractions within 3 weeks after the first immunotherapy dose.

Chemotherapy is permitted during the study in both groups. The decision to use chemotherapy will be made by the treating physician based on the patient's individual condition and prior treatment history.

Primary Endpoint Objective Response Rate (ORR) of lesions outside the radiotherapy field, assessed by RECIST 1.1 criteria.

Secondary Endpoints Disease Control Rate (DCR) of lesions outside the radiotherapy field. Safety profile (≥3 toxicities). ORR of lesions within the radiotherapy field. Distant metastasis rate outside the radiotherapy field. Progression-Free Survival (PFS) and Overall Survival (OS).

Safety Monitoring Adverse events and serious adverse events (SAE) will be closely monitored and reported according to the protocol. Treatment will be discontinued if predefined criteria for stopping are met.

Study Duration The study will include a screening period, a treatment period, and a follow-up period with regular assessments every 2 cycles of immunotherapy until death occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years；
2. Patients with recurrent/metastatic HER2-negative breast cancer；
3. Patients who have previously received standard treatment regimens for recurrent/metastatic breast cancer；
4. At least one lesion suitable for radiation therapy；
5. At least one measurable metastatic lesion outside of the radiation field, and can be monitored using the "Response Evaluation Criteria in Solid Tumors" (RECIST) version 1.1；
6. ECOG performance status of 0-2；
7. Signed informed consent；
8. Patients who have previously received radiation therapy may be included as long as it does not interfere with irradiation of the target lesion；

Exclusion Criteria:

1. Biliary obstruction, acute or chronic cholecystitis or cholangitis, or long-term biliary colic (contraindication for UDCA)；
2. Malabsorption syndrome or diseases that significantly affect gastrointestinal function; patients who have undergone total gastrectomy or resection of the proximal small intestine that may affect oral drug absorption；
3. Exclusion of patients with symptomatic brain metastases or leptomeningeal metastasis; patients with brain metastases who have been treated and stabilized (with no progression within 4 weeks) may be included, but brain metastases cannot be used as target lesions；
4. Known invasive malignancies within the past 5 years that are still progressing or require active treatment (excluding patients with basal cell carcinoma, squamous cell carcinoma of the skin, or breast ductal carcinoma in situ or cervical carcinoma in situ who have received curative treatment)；
5. Previous immune therapy resulting in grade 3 or higher adverse events； Diagnosed with immunodeficiency or receiving long-term systemic corticosteroid treatment (prednisone equivalent dose >10 mg daily) or any form of immunosuppressive therapy within 7 days before the first dose of study treatment；
6. Active autoimmune diseases requiring systemic treatment (e.g., using disease-modifying drugs, corticosteroids, or immunosuppressive drugs) within the past 2 years；
7. Active infections requiring systemic treatment；
8. Known history of active tuberculosis；
9. Other significant cardiovascular diseases, including recent myocardial infarction, acute coronary syndrome, or a history of coronary artery interventions (angioplasty, stent placement, or bypass surgery) within the last 6 months; NYHA Class II-IV congestive heart failure (CHF) or a history of NYHA Class III or IV CHF；
10. Known history of human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) of lesions outside the radiotherapy field, assessed by RECIST 1.1 criteria. | From date of randomization to 4 weeks after completion of radiotherapy

SECONDARY OUTCOMES:
Disease Control Rate (DCR) of lesions outside the radiation field, assessed by RECIST 1.1 criteria | From date of randomization to 4 weeks after completion of radiotherapy
Safety: Incidence of Grade ≥3 toxicities, assessed by CTCAE 5.0 criteria | From first dose of study drug to 30 days post-treatment completion
Objective Response Rate (ORR) of lesions within the radiation field, assessed by RECIST 1.1 criteria | From date of randomization to 4 weeks after completion of radiotherapy
Overall response assessment of lesions both within and outside the radiation field, assessed by mRECIST criteria | From date of randomization to 4 weeks after completion of radiotherapy
Progression-Free Survival (PFS): Time from randomization to the first documented progression or death, whichever occurs first | From randomization to the first documented progression or death, whichever occurs first, assessed every 6 weeks up to 48 weeks post-randomization.
Overall Survival (OS): time from randomization to death from any cause | From randomization to death from any cause, assessed continuously until all patients have died (up to 5 years post-randomization).

OTHER OUTCOMES:
Circulating Tumor Cells (CTCs) Enumeration | Within 1 week before radiotherapy, within 1 week after the completion of radiotherapy
Circulating Tumor DNA (ctDNA) | Within 1 week before radiotherapy, within 1 week after the completion of radiotherapy
Peripheral Blood Mononuclear Cell (PBMC) Immune Composition | Within 1 week before radiotherapy, within 1 week after the completion of radiotherapy
Whole Blood Immune Factor Profiling | Within 1 week before radiotherapy, within 1 week after the completion of radiotherapy